CLINICAL TRIAL: NCT05446181
Title: Accumulation of Chloride Intracellular Channel 1 (CLIC1) Protein in Circulating Monocyte in Elderly Patients Presenting Postoperative Delirium and Its Predictable Role of Postoperative Delirium
Brief Title: CLIC1 in Patients Presenting PD
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, principle investigator, Seoul National University Bundang Hospital
Other Study IDs: B-2109-706-302
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hip Fractures; Hip Disease
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Old with perioperative delirium
  Interventions: Behavioral: Perioperative delirium; Procedure: Hip surgery
- Old without perioperative delirium
  Interventions: Procedure: Hip surgery

INTERVENTIONS:
Behavioral: Perioperative delirium — Perioperative delirium
  Groups: Old with perioperative delirium
Procedure: Hip surgery — Orthopedic hip joint surgery under spinal anesthesia

SUMMARY:
In this study, mononuclear cells, particularly monocytes, were collected from the peripheral blood of elderly patients who underwent orthopedic hip surgery under spinal anesthesia. We then observe the accumulation of chloride intracellular channel 1 (CLIC1), particularly the characteristic accumulation morphology and its function. The purpose of this study is to compare whether there is a difference in the degree and form of cytoplasmic CLIC1 accumulation between the elderly group with postoperative delirium (PD) and the elderly group without postoperative delirium. We'll also confirm whether this is appropriate as a predictor of postoperative delirium. In addition, we will establish a control group for the non-elderly group to check the difference due to aging itself.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients aged 65 years or older who are scheduled to undergo surgery for an orthopedic hip fracture under spinal anesthesia

Exclusion Criteria:

* Patients who are unconscious
* Patients who are unable to communicate
* Alzheimer
* Parkinson Disease
* Conversion to general anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing hip joint surgery are divided into the PD group or non-PD group
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
expression pattern of CLIC1 protein | Immediate after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No